CLINICAL TRIAL: NCT00290628
Title: Transplantation of Umbilical Cord Blood From Related and Unrelated Donors
Brief Title: Donor Umbilical Cord Blood Transplant in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced with another study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 2000LS017; UMN-MT1999-28
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Chronic Myeloproliferative Disorders; Diamond-blackfan Anemia; Fanconi Anemia; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Diamond-Blackfan anemia; Fanconi anemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Anemia, Diamond-Blackfan; Fanconi Anemia; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Filgrastim; Melphalan; Methylprednisolone; Mycophenolic Acid; Radiotherapy; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: filgrastim
Drug: melphalan
Drug: methylprednisolone
Drug: mycophenolate mofetil
Procedure: radiation therapy
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related or unrelated donor, that do not exactly match the patient's blood, are infused into the patient they may help the patient's bone marrow to make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This clinical trial is studying how well donor umbilical cord blood transplant works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the engraftment potential of umbilical cord blood (UCB) in patients with hematological cancers.
* Determine the safety of UCB transplantation in these patients.

Secondary

* Determine the rate of neutrophil and platelet recovery and the completeness of donor cell engraftment.
* Determine the incidence and severity of acute and chronic graft-versus-host disease.
* Determine the incidence of relapse in patients with malignant disease.
* Determine the probabilities of survival and event-free survival (EFS) at 1 and 2 years after UCB transplantation.

OUTLINE: Patients are stratified according to degree of HLA disparity (0-1 vs 2-3 disparities between donor and recipient), donor type (related vs unrelated), and the basis of cell dose (< 2 vs ≥ 2 x 10^7 nucleated cells/kg recipient body weight). Patients are assigned to 1 of 4 treatment groups according to disease*.

NOTE: *Patients with acute lymphocytic leukemia (ALL), secondary acute myeloid leukemia (AML), severe combined immunodeficiency, familial erythrophagocytic lymphohistiocytosis (FEL)/viral-associated hemophagocytic syndrome (VAHS), inborn errors of metabolism, aplastic anemia, Fanconi's anemia, or Diamond-Blackfan anemia who have an unrelated umbilical cord blood donor may proceed directly to transplantation.

* Preparative regimen:

  * Group 1 (patients with chronic myelogenous leukemia, AML, myelodysplastic syndromes, or ALL): Patients receive cyclophosphamide IV once daily on days -7 and -6. Patients then undergo total-body irradiation (TBI) twice daily on days -4 to -1. Patients undergoing unrelated allogeneic umbilical cord blood transplantation (UCBT) also receive methylprednisone IV and anti-thymocyte globulin (ATG) IV twice daily on days -2 and -1.
  * Group 2 (patients with infant leukemia): Patients receive busulfan orally or IV four times daily on days -9 to -6 and melphalan IV once daily on days -4 to -2. Patients undergoing unrelated allogeneic UCBT also receive methylprednisolone IV and ATG IV twice daily on days -2 and -1.
  * Group 3 (patients with inborn errors of metabolism): Patients receive busulfan orally or IV four times daily on days -9 to -6 and cyclophosphamide IV once daily on days -5 to -2. Patients undergoing unrelated allogeneic UCBT also receive methylprednisolone IV and ATG IV twice daily on days -2 and -1.
  * Group 4 (patients with aplastic anemia): Patients receive cyclophosphamide IV once daily on days -6 to -3 and ATG IV twice daily on days -5 and -3. Patients then undergo TBI once on day -2.
* Allogeneic UCBT: Patients undergo UCBT on day 0. Patients with inborn errors of metabolism receive methylprednisolone IV before and after UCBT on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive 1 of the following regimens:

  * Related donor UCBT: Patients receive cyclosporine IV over 2 hours or orally beginning on day -3 and continuing until day 60.
  * Unrelated donor UCBT and myeloablative preparative regimen: Patients receive cyclosporine orally or IV over 2 hours twice daily beginning on day -3 and continuing until day 180. Patients also receive methylprednisolone IV twice daily on days 5-19.
  * Unrelated donor UCBT and nonmyeloablative preparative regimen: Patients receive cyclosporine IV over 2 hours or orally twice daily beginning on day -3 and continuing until day 180. Patients also receive mycophenolate mofetil IV or orally beginning on day 5 and continuing until day 30 or 7 days after active GVHD is controlled.

All patients receive filgrastim (G-CSF) IV beginning on day 1 and continuing until blood counts recover.

Patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Leukemia including, but not limited to, the following subtypes:

    * Chronic myelogenous leukemia
    * Acute myeloid leukemia (primary or secondary)
    * Acute lymphoblastic leukemia
  * Lymphoma
  * Myelodysplastic syndrome
  * Aplastic anemia
  * Fanconi's anemia
  * Diamond-Blackfan anemia
  * Inborn errors of metabolism (e.g., Hurler syndrome, Maroteaux-Lamy syndrome, myelodysplastic syndrome VI, metachromatic leukodystrophy, adrenoleukodystrophy, and globoid cell leukodystrophy)
  * Immune deficiency disorders
* Patients must meet the eligibility requirements outlined in currently active treatment protocols of the University of Minnesota Bone Marrow Transplant Program
* HLA-identical or 1, 2, or 3 antigen mismatched umbilical cord blood (UCB) donor with at least one DRB1 match available

  * Unrelated or related donor
  * UCB specimen must contain ≥ 2.0 x 10^7 nucleated cells/kg patient body weight

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* No active infection
* No history of HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 1999-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Wagner, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States